CLINICAL TRIAL: NCT03993366
Title: A Preliminary Pilot Study to Assess Insulin-plus-Pramlintide Closed-loop Delivery System in Pump Treated Patients With Type 1 Diabetes Mellitus
Brief Title: Pramlintide and Fiasp Closed-Loop With a Simple Meal Announcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-4947
Record Dates: First submitted 2019-03-11; First posted 2019-06-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; artificial pancreas; pramlintide; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study is a randomized, 2-way, crossover trial assessing:
  i. Fiasp-alone closed-loop system with full carbohydrate counting ii. Fiasp-plus-Pramlintide closed-loop system with simple meal announcement in regulating glucose levels in patients with type 1 diabetes, over a period of 24h in an inpatient setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Meal Announcement (Experimental): Before every meal, the meal will be simply announced to the algorithm by a member of the study team. Meal bolus computation will be independent of the carbohydrate content of the meal.
  Interventions: Combination Product: Fiasp+Pramlintide Closed-Loop System
- Full Carbohydrate counting (Active Comparator): The carbohydrate content of the meal selected by the participant will be entered into the dosing algorithm by a member of the study team at the onset of the meal to compute the insulin prandial bolus.
  Interventions: Device: Fiasp Closed-Loop System

INTERVENTIONS:
Combination Product: Fiasp+Pramlintide Closed-Loop System — Closed-loop insulin delivery with Fiasp insulin and pramlintide
  Arms: Simple Meal Announcement
Device: Fiasp Closed-Loop System — Closed-loop insulin delivery with Fiasp insulin alone
  Arms: Full Carbohydrate counting

SUMMARY:
The aim of this pilot study is to generate preliminary data of (i) Fiasp-plus-Pramlintide closed-loop system with a simple meal announcement, compared to (ii) Fiasp-alone closed-loop system with full carbohydrate counting, in preparation for an outpatient study over two weeks

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 12 years of age.
2. Clinical diagnosis of type 1 diabetes for at least 12 months according to the Diabetes Canada Clinical Practice Guidelines Expert Committee diagnostic criteria.
3. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
4. Insulin pump therapy for at least 6 months.
5. HbA1c ≤ 12%.

Exclusion Criteria:

1. Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2 (Sodium-glucose Cotransporter-2), GLP-1 (glucagon-like peptide 1), Metformin, Acarbose, etc.…).
2. Current use of glucocorticoid medication.
3. Use of medication that alters gastrointestinal motility.
4. Planned or ongoing pregnancy.
5. Breastfeeding individuals.
6. Severe hypoglycemic episode within one month of admission.
7. Severe diabetes keto-acidosis episode within one month of admission.
8. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
9. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
10. Known hypersensitivity to any of the study drugs or their excipients.
11. Individuals with hypoglycemia unawareness.
12. Individuals with confirmed gastroparesis.
13. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
14. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Study Discontinuation/Withdrawal

1. Failure to comply with the protocol.
2. Pregnancy.
3. After an event which the PI believes it is not in the best interest for the patient to continue the trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Time in target | 24 hours
  Time spent in target range (between 4.0 mmol/L and 10 mmol/L)
Time in hypoglycemia | 24 hours
  Time spent in hypoglycemic range (below 4.0 mmol/L)
Time in hyperglycemia | 24 hours
  Time spent in hyperglycemic range (above 10.0 mmol/L)

OTHER OUTCOMES:
Hypoglycemia treatment | 24 hrs
  Number of participants experiencing hypoglycemia requiring oral treatment
Hypoglycemia treatment | During the night of the 24 hour intervention (11pm-7am)
  Number of participants experiencing hypoglycemia requiring oral treatment
Hypoglycemia treatment | During the day of the 24 hour intervention (7am-11pm)
  Number of participants experiencing hypoglycemia requiring oral treatment
Gastrointestinal symptoms | 24 hours
  Presence of gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided